CLINICAL TRIAL: NCT06980077
Title: UCLA L-11: A Phase II Trial of Ivonescimab for Previously Treated Thymic Carcinoma
Brief Title: Ivonescimab for the Treatment of Thymic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-6289; NCI-2025-03012 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-05

CONDITIONS: Thymus Carcinoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (ivonescimab) (Experimental): Patients receive ivonescimab IV over 60-120 minutes on day 1 of each cycle. Cycles repeat Q3W for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and collection of blood and urine samples throughout the study. Patients may undergo MRI throughout the study if indicated and may optionally undergo a biopsy at the end of treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ivonescimab; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Ivonescimab — Given IV
  Other Names: AK 112; AK-112; AK112; Anti-PD-1/Anti-VEGF Bispecific Antibody AK112; Anti-PD-1/VEGF Bispecific Antibody AK112; PD-1/VEGF Bispecific Antibody AK112; SMT 112; SMT-112; SMT112
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well ivonescimab works in treating patients with thymic carcinoma. Immunotherapy with monoclonal antibodies, such as ivonescimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure anti-tumor effect of ivonescimab for thymic carcinoma (TC) as measured by overall response rate (ORR), which is defined as complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

II. Assess the safety and tolerability of ivonescimab for thymic carcinoma.

SECONDARY OBJECTIVE:

I. To evaluate the efficacy of ivonescimab as measured progression free survival (PFS), duration of response (DOR), time to response (TTR) and overall survival (OS).

EXPLORATORY OBJECTIVE:

I. Assess potential biomarkers associated with response from liquid biopsies and archival tissue samples.

OUTLINE:

Patients receive ivonescimab intravenously (IV) over 60-120 minutes on day 1 of each cycle. Cycles repeat once every 3 weeks (Q3W) for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and collection of blood and urine samples throughout the study. Patients may undergo magnetic resonance imaging (MRI) throughout the study if indicated and may optionally undergo a biopsy at the end of treatment.

After completion of study treatment, patients are followed up every 6 weeks through week 24, and then every 12 weeks thereafter for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age and willing and able to provide informed consent
* Cytologically or histologically confirmed thymic carcinoma, which is incurable
* Received prior systemic therapy for thymic carcinoma, or is ineligible for or refuses other therapies
* Measurable disease, as per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
* Platelets ≥ 100 × 10^9/L
* Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCl) ≥ 50 mL/min (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl)

  * Estimated glomerular filtration rate (eGFR) value ≥ 50 mL/min for participants with creatinine levels > 1.5 x institutional ULN
  * Creatinine clearance may be calculated using the Cockcroft-Gault formula or estimated glomerular filtration rate (eGFR) may be calculated using the Modification of Diet in Renal Disease (MDRD) GFR equation
* Urine dipstick protein ˂ 2+ OR 24 hour urine protein quantification ˂ 1.0 g
* Serum total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x ULN OR ≤ 5 x ULN for participants with liver metastases
* Albumin ≥ 2.5 g/dL
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy, and then only as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy, and then only as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female participants of childbearing potential must have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the participant to be eligible. Female participants must agree to use a highly effective method of contraception from the beginning of screening until 120 days after the last dose of the ivonescimab, or be of non-childbearing potential. Non-childbearing potential is defined as follows (by other than medical reasons):

  * ≥ 45 years of age and has not had menses for > 2 years,
  * Participants who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation, or
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation
* Unsterilized male patients having sex with a female partner of childbearing potential, or a pregnant or breastfeeding partner must agree to use barrier contraception (male condom) for the duration of the treatment period until 120 days after the last dose of ivonescimab. Male patients with female partners of childbearing potential must have the female partner agree to use at least 1 form of highly effective contraception for the duration of the treatment period until 120 days after the last dose of ivonescimab
* Male and female participants must agree not to donate sperm or eggs, respectively, from the first study-drug treatment through 120 days after the last study drug treatment
* Female participants must agree to not breastfeed during the study or for 120 days after the last dose of study treatment

Exclusion Criteria:

* Prior treatment with an immune checkpoint inhibitor targeted PD-1 or PD-L1. Prior treatment with VEGF inhibitor is allowed
* Concurrent enrollment in another clinical study, unless enrolled only in the follow-up period or an observational study
* Any chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment in the prior 3 weeks or within 5 half-lives of the medication, whichever is shorter. Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable
* Thoracic radiation of ≥ 30 Gy within 3 months. Other radiation within 3 weeks with the following exceptions: (a) Stereotactic, palliative radiation for bone metastases is acceptable without a washout; (b) Stereotactic brain radiation for asymptomatic brain metastases is acceptable with a 7 day washout
* Use of any investigational anticancer therapy received within 21 days prior to the first dose of study drug
* Has not recovered (recovery is defined as National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE version (v)5.0] grade ≤ 1) from the acute toxicities of previous therapy, except treatment-related alopecia, sensory neuropathy, or laboratory abnormalities otherwise meeting the inclusion requirements stated in the inclusion criterion. Other grade 2 or less toxicities not constituting a safety risk based on the investigator's judgment are acceptable
* The patient has a known allergy/history of hypersensitivity reaction to any of the treatment components or any other contraindication to one of the administered treatments
* Active autoimmune condition currently requiring systemic immune suppressive therapy
* Positive paraneoplastic serologies, including binding, blocking and modulating antibodies to acetylcholine receptor (AChR)

  * If known muscle-specific kinase (MuSK) antibodies positive then excluded, otherwise additional testing not required
* Major surgical procedures or serious trauma within 4 weeks prior to randomization, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to randomization
* Poorly controlled hypertension with repeated systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy
* Presence of angina or active cardiac ischemia, uncontrolled congestive heart failure of current ≥ class III as defined by the New York Heart Association, or unstable cardiac arrhythmia (e.g., clinically stable atrial fibrillation is permitted)
* The patient has experienced myocardial infarction within 6 months prior to study enrollment
* History of arterial or venous thrombosis or thromboembolism within 6 months prior to study enrollment. Patients with a history of venous thromboembolism beyond 6 months prior to study enrollment can be enrolled if they are appropriately anticoagulated
* Imaging during the screening period shows that the tumor surrounds important blood vessels or has obvious necrosis and/or cavitation, and the investigator determines that entering the study is a bleeding or fistula risk. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted
* The patient has any ongoing or active infection requiring the use of parenteral anti-microbial agents, or grade > 2 by NCI CTCAE (v5.0) within 14 days prior to enrollment. Patient with a history of HIV with an undetectable viral load and cluster of differentiation 4 (CD4) count over 200 are eligible. Patients with a history of hepatitis B or hepatitis C, an undetectable viral load, and liver function test (LFT) testing which meets criteria for the study are eligible
* The patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 210 days after the last dose of trial treatment
* Progressive or symptomatic brain metastases. Brain metastases that have been radiated, are asymptomatic, and on a stable or decreasing dose of steroids are allowed. Leptomeningeal disease is excluded
* History of another cancer within 2 years of study initiation, with the exception of fully treated cancers unlikely to affect the assessment of the study treatment safety or efficacy including early stage breast, prostate, bladder, non-melanomatous skin, thyroid, cervical, or endometrial cancer
* History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to randomization, including but not limited to:

  * Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots)

    * Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed
  * Nasal bleeding/epistaxis (bloody nasal discharge is allowed)
* Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to randomization is not allowed. The use of full-dose anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits according to the medical standard of the enrolling institution. History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before randomization
* History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to randomization
* Active autoimmune or lung disease requiring systemic therapy (eg, with disease modifying drugs, prednisone > 10 mg daily or equivalent, immunosuppressant therapy) within 2 years prior to randomization, however the following will be allowed:

  * Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted.
  * Intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections is permitted
* Has pre-existing peripheral neuropathy that is ≥ grade 2 by CTCAE version 5
* Uncontrolled pleural effusions, pericardial effusions, or ascites that is clinically symptomatic

  * Patients managed with indwelling catheters (eg, PleurX) are allowed
* History of non-infectious pneumonia requiring systemic corticosteroids, or current interstitial lung disease
* Active or prior history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Known history of human immunodeficiency virus (HIV) whose viral load is not controlled
* Current use of systemic corticosteroids (> 10 mg daily prednisone or equivalent)
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Live vaccine or live attenuated vaccine within 4 weeks prior to planned randomization, or if scheduled to receive a live vaccine or live attenuated vaccine during the study period. Inactivated vaccines are permitted
* Participants must not be considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Patient unwilling or unable to comply with the protocol
* Any condition that, in the opinion of the investigator or sponsor, would interfere with evaluation of the investigational product or interpretation of subject safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-06-17 (Estimated); Study Completion 2028-06-17 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 1 year
  ORR is defined as complete response or partial response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. The ORR estimate and its associated 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Progression free survival | From trial initiation to cancer progression or death due to any cause, assessed up to 1 year
  Cancer progression will be determined per RECIST 1.1.
Duration of response | From documentation of tumor response to disease progression, assessed up to 1 year
Time to response | From treatment initiation until documentation of tumor response, assessed up to 1 year
Overall survival | From randomization to death by any cause, assessed up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Goldman, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States